CLINICAL TRIAL: NCT07324473
Title: Ivarmacitinib Combined With Camrelizumab and Apatinib for Unresectable Advanced Hepatocellular Carcinoma With Acquired Resistance to Immune Checkpoint Therapy: A Single-Arm Exploratory Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Gu Jinyang, Director of Hepatobiliary and Pancreatic Surgery Department, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-817-01
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinomas; Resistance to Immunotherapy; Immunomodulation; Drug Repurposing
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental treatment group (Experimental)
  Interventions: Drug: The triple-therapy strategy of Ivarmacitinib, Apatinib, and Camrelizumab

INTERVENTIONS:
Drug: The triple-therapy strategy of Ivarmacitinib, Apatinib, and Camrelizumab — All enrolled patients will receive triple therapy consisting of Ivarmacitinib (4mg, orally, qd, starting immediately upon enrollment completion) + Apatinib (250mg, orally, qd, starting on day 8 after the initiation of Ivarmacitinib) + Camrelizumab (200mg, intravenous infusion, q3w, starting on day 8 after the initiation of Ivarmacitinib). Treatment will continue until disease progression, unacceptable toxicity, or for up to 2 years.

SUMMARY:
Background： Hepatocellular carcinoma (HCC) stands as a formidable global health challenge. It ranks as the sixth most common malignant solid tumor worldwide and the third leading cause of cancer-related mortality. The disease is characterized by its insidious onset, rapid progression, and high recurrence rates, contributing to a dismal 5-year survival rate of approximately 18%. A critical factor in this poor prognosis is that nearly 57% of patients are diagnosed at an advanced stage, where curative surgical resection is no longer feasible. For these patients with unresectable advanced HCC (uHCC), effective systemic therapies are paramount to extend survival and improve quality of life.

The advent of immunotherapy, particularly immune checkpoint inhibitors (ICIs) targeting the PD-1/PD-L1 axis, has revolutionized the treatment landscape for numerous advanced cancers, including uHCC. These agents work by blocking the inhibitory signals that tumor cells exploit to evade immune surveillance, thereby reactivating cytotoxic T cells to attack the cancer.

However, the clinical benefit of ICI-based therapies is not universal. A substantial proportion of patients-estimated between 15% to 40%-derive limited or no benefit. Primary resistance is defined as a lack of initial response, while acquired resistance refers to disease progression after an initial period of clinical benefit. There is no established, evidence-based standard of therapy for uHCC patients who progress following first-line ICI combination therapy, highlighting an urgent need for novel therapeutic approaches.

The mechanisms underlying acquired resistance to ICIs are multifaceted and intricately linked to dynamic remodeling of the tumor immune microenvironment (TME). Several key pathways contribute:

1. Loss of Tumor Immunogenicity: Immune editing during treatment can select for tumor cell clones with low neoantigen expression, making them less visible to the immune system.
2. Immune Suppressive Cell Infiltration: The TME in resistant tumors often exhibits an accumulation of immunosuppressive cell populations, including regulatory T cells (Tregs), tumor-associated macrophages (TAMs), and myeloid-derived suppressor cells (MDSCs). These cells create a profoundly inhibitory milieu that dampens anti-tumor T cell function.
3. T Cell Exhaustion: Persistent antigen exposure leads to a state of CD8⁺ T cell exhaustion, rendering them dysfunctional.

These interconnected mechanisms collectively foster an immunosuppressive TME that allows tumors to evade ongoing immune attack, underscoring the need for combination strategies that can reshape the TME and re-sensitize tumors to immunotherapy.

The JAK-STAT pathway serves as a critical signaling hub for numerous cytokines and growth factors, playing a pivotal dual role in immunity and inflammation. In the context of HCC and ICI resistance, its activation is particularly relevant:

1. Pathway Activation in HCC: The JAK/STAT pathway is ubiquitously activated in both primary and recurrent HCC tumors and contributes to the proliferation and survival of tumor-initiating cells.
2. Driver of an Immunosuppressive TME: Hyperactivation of this pathway, often via cytokines like IL-6, promotes the recruitment and activation of immunosuppressive MDSCs and M2-polarized TAMs. It also contributes to T cell exhaustion.
3. Preclinical and Clinical Proof-of-Concept: In preclinical models, JAK/STAT inhibition has been shown to reduce MDSC infiltration and restore T cell function. Most compellingly, recent clinical studies in other cancer types published in high-impact journals like Science (2024) have demonstrated that adding a JAK inhibitor to PD-1 blockade can re-sensitize tumors and yield significant clinical responses in patients who had developed resistance to immunotherapy alone

Purpose:

This single-arm, exploratory clinical study aims to evaluate the efficacy and safety of Ivarmacitinib (a selective JAK1 inhibitor) combined with Camrelizumab (anti-PD-1) and Apatinib (anti-VEGFR2) in patients with advanced unresectable HCC who have progressed after first-line ICI-based combination therapy.

Methods:

This study plans to enroll 65 patients with advanced unresectable hepatocellular carcinoma (unresectable BCLC stage B or stage C) who have been clinically or pathologically diagnosed, have previously received at least 4 cycles of guideline-recommended first-line targeted therapy combined with PD-1/PD-L1 immunotherapy, achieved a partial response, but subsequently experienced disease progression confirmed by RECIST 1.1 criteria after at least 4 cycles (indicating acquired resistance).

All enrolled patients will receive triple therapy consisting of Ivarmacitinib + Apatinib + Camrelizumab. Treatment will continue until disease progression, unacceptable toxicity, or for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of hepatocellular carcinoma, confirmed either by clinical diagnosis (per the Chinese Guidelines for the Diagnosis and Treatment of Primary Liver Cancer [2022 Edition]) or by pathological diagnosis.
2. Patients classified as Barcelona Clinic Liver Cancer (BCLC) stage B and assessed by the responsible hepatobiliary surgeon as unsuitable for radical resection, or patients with BCLC stage C disease.
3. Patients with unresectable hepatocellular carcinoma who have developed secondary (acquired) drug resistance. This is defined as having received at least 4 cycles of a first-line targeted therapy combined with immunotherapy regimen recommended by guidelines . Eligible prior regimens include specified combinations (e.g., Camrelizumab + Apatinib; Atezolizumab + Bevacizumab; Sintilimab + Bevacizumab) or other guideline-recommended first-line targeted agents (Donafenib, Lenvatinib, Sorafenib, Cabozantinib, Regorafenib) combined with first-line immunotherapy (Tislelizumab, Durvalumab, Pembrolizumab). Furthermore, patients must have achieved a partial response in the primary lesion but subsequently experienced disease progression after the 4th immunotherapy cycle, as confirmed per RECIST 1.1 criteria (including increase in size of primary lesion, or emergence of new lesions/metastases).
4. At least one measurable lesion according to RECIST 1.1 criteria (target lesion with longest diameter ≥ 10 mm, or lymph node with short axis ≥ 15 mm).
5. Anticipated life expectancy > 3 months.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
7. Adequate organ and bone marrow function, as evidenced by the following laboratory values within 7 days prior ： (1)Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L in the absence of granulocyte colony-stimulating factor support within the last 14 days; (2)Platelets ≥ 60 × 10⁹/L without transfusion within the last 14 days; (3)Hemoglobin > 9 g/dL without transfusion or erythropoietin use within the last 14 days; (4)Total bilirubin ≤ 2 × upper limit of normal (ULN); (5)Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; (6)Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min; (7)Adequate coagulation function, defined as an International Normalized Ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; (8)Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, study participants may still be enrolled if total T3 (or free T3) and free T4 are within the normal range; (9)Myocardial enzyme profile within normal limits (isolated laboratory abnormalities judged by the investigator as clinically insignificant are also permitted);
8. For female study participants of childbearing potential, a negative urine or serum pregnancy test must be obtained within 3 days prior to the first dose of study drug (Cycle 1, Day 1). If the urine pregnancy test result is not confirmatory, a serum pregnancy test is required. A female not of childbearing potential is defined as being postmenopausal for at least 1 year, or surgically sterilized, or having undergone a hysterectomy.

Exclusion Criteria:

* 1. Diagnosis of malignancies other than liver cancer within 5 years prior to the first dose.

  2. Intrahepatic or extrahepatic cholangiocarcinoma, combined hepatocellular-cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, fibrolamellar HCC, ampullary tumors, or other biliary tract malignancies.

  3. Prior treatment with any JAK inhibitor.

  4. Patients with pleural effusion, ascites, or pericardial effusion requiring drainage, who are clinically assessed as unable to tolerate the study treatment.

  5. History of esophageal or gastric variceal bleeding due to portal hypertension within 6 months prior to the first dose; or current imaging (contrast-enhanced CT or MRI) confirming significant esophageal or gastric varices.

  6. History of severe bleeding tendency or coagulopathy; clinically significant hemorrhagic symptoms within 1 month prior to the first dose (including but not limited to gastrointestinal bleeding, hemoptysis, epistaxis)

  7. History of myocarditis, cardiomyopathy, or malignant arrhythmia

  8. History of immunodeficiency; positive HIV antibody test; current long-term use of systemic corticosteroids or other immunosuppressants; active autoimmune disease requiring systemic treatment within the past two years.

  9. Known active tuberculosis (TB).

  10. Known active syphilis infection.

  11. Administration of a live or live-attenuated vaccine within 30 days prior to the first dose.

  12. History of mental illness, drug abuse, alcoholism, or substance abuse.

  13. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  Tumor imaging assessments (RECIST 1.1) will be performed every 6 weeks within the first year after treatment initiation and every 9 weeks thereafter.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 years
  every 6 weeks within the first year after treatment initiation and every 9 weeks thereafter.
Progression-Free Survival (PFS) | 2 years
  every 6 weeks within the first year after treatment initiation and every 9 weeks thereafter.
Overall Survival (OS) | 2 years
  Overall Survival (OS) will be assessed from the date of first study treatment until the date of death from any cause.
Adverse Events | 2 years
  Count of adverse events by grade was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to adverse event. Serious is defined as any grade 3 or higher adverse event. Toxicity is defined as any study drug-related Grade 3 or higher adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China